CLINICAL TRIAL: NCT02374021
Title: Treatments Against RA and Effect on FDG-PET/CT (The TARGET Trial)
Brief Title: Treatments Against RA and Effect on FDG-PET/CT
Acronym: TARGET
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Columbia University (Other)
Responsible Party: Principal Investigator, Daniel H. Solomon, M.D.,MPH, Chief, Section of Clinical Sciences, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2014P002747
Record Dates: First submitted 2015-02-11; First posted 2015-02-27 (Estimated); Results first posted 2022-10-26 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: Arthritis, Rheumatoid
Keywords: rheumatoid arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Methotrexate; Sulfasalazine; Hydroxychloroquine; Etanercept; Adalimumab

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Triple therapy (MTX+SSZ+HCQ) (Active Comparator): Sulfasalazine (SSZ) 1 g bid and hydroxychloroquine (HCQ) 200 mg twice daily, not to exceed 6.5mg/kg HCQ (in addition to concomitant methotrexate [MTX]).
  Interventions: Drug: Methotrexate; Drug: Sulfasalazine; Drug: Hydroxychloroquine
- TNF inhibitor (etanercept or adalimumab) (Active Comparator): etanercept 50 mg subcutaneously weekly or adalimumab 40 mg subcutaneously every other week (in addition to concomitant methotrexate, plus hydroxychloroquine, for subjects who were taking this at screening). Biologic treatment will be assigned randomly.
  Interventions: Drug: Methotrexate; Drug: Etanercept; Drug: Adalimumab

INTERVENTIONS:
Drug: Methotrexate — Subjects entering trial will continue on MTX dose of at least 15mg MTX/week. At the discretion of the treating rheumatologist, may be switched to SQ route.
  Other Names: Rheumatrex
Drug: Sulfasalazine — 1 gm bid
  Other Names: Azulfidine
  Arms: Triple therapy (MTX+SSZ+HCQ)
Drug: Hydroxychloroquine — 200 mg twice daily, not to exceed 6.5mg/kg
  Other Names: Plaquenil
  Arms: Triple therapy (MTX+SSZ+HCQ)
Drug: Etanercept — 50 mg SC weekly
  Other Names: enbrel
  Arms: TNF inhibitor (etanercept or adalimumab)
Drug: Adalimumab — 40 mg SQ every other week
  Other Names: Humira
  Arms: TNF inhibitor (etanercept or adalimumab)

SUMMARY:
In a randomized controlled clinical trial, investigators will compare the effects on [18F]-fluorodeoxyglucose positron emission tomography-computed tomography (FDG PET/CT) from two treatment regimens in rheumatoid arthritis (RA) patients deemed methotrexate inadequate responders (MTX-IRs). Two common RA treatments will be compared: triple therapy (sulfasalazine, methotrexate, and hydroxychloroquine) versus tumor necrosis factor (TNF) inhibitor (etanercept or adalimumab, plus background methotrexate for all subjects and hydroxychloroquine for subjects who were taking this at screening).

DETAILED DESCRIPTION:
Consenting subjects will be screened for eligibility and randomized to a treatment arm. Subjects will be randomized to a treatment arm with either synthetic disease-modifying antirheumatic drugs (DMARDs) [triple therapy: sulfasalazine, methotrexate, and hydroxychloroquine] or biologic DMARDs [etanercept or adalimumab, plus background methotrexate for all subjects and hydroxychloroquine for subjects who were taking this at screening].

Once randomized, a baseline visit will be conducted with each subject. Baseline data collection includes questionnaires, disease activity score, and the first FDG-PET/CT imaging. After the baseline at week 0, subjects will visit with their rheumatologist at weeks 6, 12, 18, and 24 for safety labs and further collection of disease activity scores and questionnaires. The second FDG-PET/CT will be performed at week 24. Blood specimens will be collected at weeks 0, 6, 18, and 24 for bioassays. Subject participation will end after the week 24 visit.

Patients and care providers will be unblinded. The FDG-PET/CT image readers will be blinded to treatment arm as well as timepoint of image acquisition.

ELIGIBILITY:
Inclusion Criteria:

* Fulfill American College of Rheumatology/European League Against Rheumatism 2010 criteria for RA
* Men ≥ 45 years and women ≥ 50 years
* MTX monotherapy for ≥ 8 weeks at ≥ 15mg weekly or ≥ 7.5 mg weekly with a documented intolerance to higher doses
* No non-biologic DMARDs in preceding two months (other than MTX and HCQ)
* Disease Activity Score-28 > 3.2
* Able to sign informed consent

Exclusion Criteria:

* Use of biologic DMARD within the past 6 months or use of rituximab ever
* Current use of >10mg per day of prednisone
* Use of a high-intensity statin lipid lowering drug or PCSK9 inhibitor in the past 12 months
* Prior patient reported, physician diagnosed clinical cardiovascular (CV) event
* Insulin-dependent or uncontrolled diabetes mellitus (DM)
* Systemic lupus erythematosus (SLE) or other autoimmune and chronic inflammatory diseases (i.e. inflammatory bowel disease, sarcoidosis)
* Cancer treated in the last 5 years (except basal and squamous cell) or any lymphoma or melanoma
* Known pregnancy, HIV, Hepatitis B Virus, Hepatitis C Virus, active (or untreated latent) tuberculosis
* Baseline: liver, renal or blood count abnormalities, Glucose-6-phosphate dehydrogenase (G6PD) deficiency
* Known sulfa allergy, macular disease or hypersensitivity to treatments; known demyelinating disease; uncompensated Congestive Heart Failure (CHF)
* Intra-articular injection within the 4 weeks prior to baseline FDG PET/CT
* 2 or more high dose radiation scans in the past year (CT scan with contrast, angiogram, SPECT nuclear medicine scan, myocardial/cardiac perfusion scan)

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2016-07; Primary Completion 2021-05 (Actual); Study Completion 2021-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Solomon, Principal Investigator — Brigham and Women's Hospital
Locations (31):
- United States (31):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Loma Linda University Clinical Trial Center, Loma Linda, California
  - David Geffen School of Medicine at UCLA, Los Angeles, California
  - Brigid Freyne, MD Inc., Murrieta, California
  - Desert Medical Advances, Palm Desert, California
  - University of California San Francisco, San Francisco, California
  - Nazanin Firooz MD, Inc., West Hills, California
  - Robert W. Levin, MD, PA, Clearwater, Florida
  - IRIS Research and Development, Plantation, Florida
  - Southwest Florida Clinical Research Center, Tampa, Florida
  - University of Kentucky, Lexington, Kentucky
  - The Center for Rheumatology and Bone Research, Wheaton, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Washington University Medical Center, St Louis, Missouri
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Northwell Health, Great Neck, New York
  - New York University School of Medicine, New York, New York
  - Mount Sinai- Icahn School of Medicine, New York, New York
  - Columbia University Medical Center, New York, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - Altoona Research Center, Duncansville, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Metroplex Clinical Research Center, Dallas, Texas
  - University of Texas Health Science Center at Houston, Houston, Texas
  - Baylor Scott & White Medical Center- Temple, Temple, Texas
  - Seattle Rheumatology Associates, Seattle, Washington

REFERENCES:
- [Derived] Liao KP, Rist P, Giles J, Santacroce L, Connelly MA, Glynn RJ, Ridker P, Tawakol A, Bathon J, Solomon DH. Impact of RA treatment strategies on lipids and vascular inflammation in rheumatoid arthritis: a secondary analysis of the TARGET randomized active comparator trial. Arthritis Res Ther. 2024 Jun 24;26(1):123. doi: 10.1186/s13075-024-03352-3. PMID 38915065
- [Derived] Solomon DH, Giles JT, Liao KP, Ridker PM, Rist PM, Glynn RJ, Broderick R, Lu F, Murray MT, Vanni K, Santacroce LM, Abohashem S, Robson PM, Fayad Z, Mani V, Tawakol A, Bathon J; TARGET Trial Consortium. Reducing cardiovascular risk with immunomodulators: a randomised active comparator trial among patients with rheumatoid arthritis. Ann Rheum Dis. 2023 Mar;82(3):324-330. doi: 10.1136/ard-2022-223302. Epub 2022 Nov 30. PMID 36450449

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Triple Therapy (MTX+SSZ+HCQ) | TNF Inhibitor (Etanercept or Adalimumab)
Started | 80 | 79
Completed | 57 | 58
Not Completed | 23 | 21
Not completed — Adverse Event | 1 | 0
Not completed — Lost to Follow-up | 3 | 2
Not completed — Physician Decision | 0 | 3
Not completed — Withdrawal by Subject | 6 | 5
Not completed — Poor Adherence | 0 | 1
Not completed — Scan protocol not followed | 0 | 1
Not completed — Poor quality scan/scan not able to be analyzed | 13 | 9

BASELINE CHARACTERISTICS:
Population: Baseline Patient Characteristics of Patients Included in Final Analyses
Groups:
- Total: Total of all reporting groups
Arm/Group | Triple Therapy (MTX+SSZ+HCQ) | TNF Inhibitor (Etanercept or Adalimumab) | Total
Number analyzed (Participants) | 57 | 58 | 115
Age, Continuous [Mean (Inter-Quartile Range); unit: years] | 59.0 [54.0 to 63.0] | 58.0 [53.0 to 66.0] | 58.0 [53.0 to 65.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 39 | 82
  Male | 14 | 19 | 33
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 16 | 15 | 31
  Not Hispanic or Latino | 41 | 43 | 84
  Unknown or Not Reported | 0 | 0 | 0
DAS28-CRP [Median (Inter-Quartile Range); unit: units on a scale] — Disease Activity Score-28 for Rheumatoid Arthritis using C-reactive protein
  The DAS28 score uses:
  * The number of swollen joints (out of the 28),
  * The number of tender joints (out of the 28),
  * The C reactive protein (CRP) or erythrocyte sedimentation rate (ESR) lab test results (value greater than zero)
  * Answers to a patient GLOBAL health assessment questionnaire (visual analog scale, 0 to 10)
  Range of the DAS-28 is 0 to 10; <2.6 represents disease remission, 2.6-3.2 represents low disease activity, >3.2-5.1 represents moderate disease activity, >5.1 represents high disease activity
  units on a scale | 4.6 [3.7 to 5.6] | 4.9 [4.0 to 5.5] | 4.8 [4.0 to 5.6]

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Vascular Inflammation as Measured by FDG-PET/CT at 6 Months
Description: The primary outcome was the change in the mean of the maximum of the target to background ratio (TBR) in the most diseased segment (MDS) of of the index vessel as measured by FDG-PET/CT scans conducted at baseline and after 24 weeks of randomized treatment allocation (MDS meanmaxTBR). The index vessel is the vessel (either aorta, left carotid, or right carotid) with the highest meanmaxTBR at baseline. Higher values indicate greater vascular inflammation.
  FDG uptake measurement: PET-CT images were batch-analyzed by an investigator blinded to the patients' clinical information. FDG uptake was evaluated within the wall of the ascending aorta and bilateral carotid arteries (as maximum and mean standardized FDG uptake value [SUVmax and SUVmean, respectively]) approximately every 5 mm on axial images. Subsequently, the target-to-background ratio (TBR) was reported (ratio of the average arterial to blood axial slice SUVmax) to correct for the blood compartment contribution.
Time Frame: 0, 6 months
Population: Participants with a FDG-PET/CT at baseline and six months for whom the primary outcome could be assessed
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Triple Therapy (MTX+SSZ+HCQ) | TNF Inhibitor (Etanercept or Adalimumab)
Number analyzed (Participants) | 57 | 58
ratio | -0.19 (0.51) | -0.24 (0.51)
Statistical Analysis 1: Comparison: Triple Therapy (MTX+SSZ+HCQ) vs TNF Inhibitor (Etanercept or Adalimumab); Test type: Superiority; p = 0.79, ANCOVA; Mean Difference (Final Values) = -0.02, 95% CI 2-sided [-0.19 to 0.15]

2. Secondary Outcome: Change From Baseline in the MDS of the Aorta
Description: The outcome was the change in the mean of the maximum of the target to background ratio (TBR) in the most diseased segment (MDS) of the aorta as measured by FDG-PET/CT scans conducted at baseline and after 24 weeks of randomized treatment allocation (MDS meanmaxTBR). Higher values indicate greater vascular inflammation.
  FDG uptake measurement: PET-CT images were batch-analyzed by an investigator blinded to the patients' clinical information. FDG uptake was evaluated within the wall of the ascending aorta and bilateral carotid arteries (as maximum and mean standardized FDG uptake value [SUVmax and SUVmean, respectively]) approximately every 5 mm on axial images. Subsequently, the target-to-background ratio (TBR) was reported (ratio of the average arterial to blood axial slice SUVmax) to correct for the blood compartment contribution.
Time Frame: 0, 6 months
Population: Participants with a FDG-PET/CT at baseline and six months for whom the outcome could be assessed
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Triple Therapy (MTX+SSZ+HCQ) | TNF Inhibitor (Etanercept or Adalimumab)
Number analyzed (Participants) | 52 | 56
Ratio | -0.17 (0.39) | -0.17 (0.52)
Statistical Analysis 1: Comparison: Triple Therapy (MTX+SSZ+HCQ) vs TNF Inhibitor (Etanercept or Adalimumab); Test type: Superiority; p = 0.05, ANCOVA; Mean Difference (Final Values) = 0.01, 95% CI 2-sided [-0.14 to 0.17]

3. Secondary Outcome: Change From Baseline in the Average TBR of the Aorta
Description: The outcome was the change in the target to background ratio (TBR) of the aorta as measured by FDG-PET/CT scans conducted at baseline and after 24 weeks of randomized treatment allocation (MDS meanmaxTBR). Higher values indicate greater vascular inflammation.
  FDG uptake measurement: PET-CT images were batch-analyzed by an investigator blinded to the patients' clinical information. FDG uptake was evaluated within the wall of the ascending aorta and bilateral carotid arteries (as maximum and mean standardized FDG uptake value [SUVmax and SUVmean, respectively]) approximately every 5 mm on axial images. Subsequently, the target-to-background ratio (TBR) was reported (ratio of the average arterial to blood axial slice SUVmax) to correct for the blood compartment contribution.
Time Frame: 0, 6 months
Population: Participants with a FDG-PET/CT at baseline and six months for whom the outcome could be assessed
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Triple Therapy (MTX+SSZ+HCQ) | TNF Inhibitor (Etanercept or Adalimumab)
Number analyzed (Participants) | 52 | 56
Ratio | -0.06 (0.34) | -0.02 (0.43)
Statistical Analysis 1: Comparison: Triple Therapy (MTX+SSZ+HCQ) vs TNF Inhibitor (Etanercept or Adalimumab); Test type: Superiority; p = 0.05, ANCOVA; Mean Difference (Final Values) = 0.03, 95% CI 2-sided [-0.11 to 0.18]

4. Secondary Outcome: Change From Baseline in the Average TBR of the Bilateral Carotids
Description: The outcome was the change in the target to background ratio (TBR) of the average of the left and right carotids as measured by FDG-PET/CT scans conducted at baseline and after 24 weeks of randomized treatment allocation (MDS meanmaxTBR). The baseline values of the left and right carotids were averaged and then the follow-up values of the left and right carotids were averaged resulting in one value at each time point. Higher values indicate greater vascular inflammation.
  FDG uptake measurement: PET-CT images were batch-analyzed by an investigator blinded to the patients' clinical information. FDG uptake was evaluated within the wall of the ascending aorta and bilateral carotid arteries (as maximum and mean standardized FDG uptake value [SUVmax and SUVmean, respectively]) approximately every 5 mm on axial images. Subsequently, the target-to-background ratio (TBR) was reported (ratio of the average arterial to blood axial slice SUVmax) to correct for the blood compartment contribution.
Time Frame: 0, 6 months
Population: Participants with a FDG-PET/CT at baseline and six months for whom the outcome could be assessed
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Triple Therapy (MTX+SSZ+HCQ) | TNF Inhibitor (Etanercept or Adalimumab)
Number analyzed (Participants) | 43 | 45
Ratio | -0.10 (0.51) | -0.06 (0.48)
Statistical Analysis 1: Comparison: Triple Therapy (MTX+SSZ+HCQ) vs TNF Inhibitor (Etanercept or Adalimumab); Test type: Superiority; p = 0.05, ANCOVA; Mean Difference (Final Values) = -0.003, 95% CI 2-sided [-0.20 to 0.19]

5. Secondary Outcome: Change From Baseline in the Average TBR of the Index Vessel
Description: The outcome was the change in the target to background ratio (TBR) in the index vessel as measured by FDG-PET/CT scans conducted at baseline and after 24 weeks of randomized treatment allocation (MDS meanmaxTBR). Higher values indicate greater vascular inflammation.
  FDG uptake measurement: PET-CT images were batch-analyzed by an investigator blinded to the patients' clinical information. FDG uptake was evaluated within the wall of the ascending aorta and bilateral carotid arteries (as maximum and mean standardized FDG uptake value [SUVmax and SUVmean, respectively]) approximately every 5 mm on axial images. Subsequently, the target-to-background ratio (TBR) was reported (ratio of the average arterial to blood axial slice SUVmax) to correct for the blood compartment contribution.
Time Frame: 0, 6 months
Population: Participants with a FDG-PET/CT at baseline and six months for whom the outcome could be assessed
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Triple Therapy (MTX+SSZ+HCQ) | TNF Inhibitor (Etanercept or Adalimumab)
Number analyzed (Participants) | 57 | 58
Ratio | -0.07 (0.47) | -0.09 (0.43)
Statistical Analysis 1: Comparison: Triple Therapy (MTX+SSZ+HCQ) vs TNF Inhibitor (Etanercept or Adalimumab); Test type: Superiority; p = 0.05, ANCOVA; Mean Difference (Final Values) = -0.01, 95% CI 2-sided [-0.17 to 0.16]

ADVERSE EVENTS:
Time Frame: 24 weeks
Arm/Group | Triple Therapy (MTX+SSZ+HCQ) | TNF Inhibitor (Etanercept or Adalimumab)
All-Cause Mortality (participants affected / at risk) | 0/80 | 0/79
Serious Adverse Events (participants affected / at risk) | 4/80 | 10/79
Other Adverse Events (participants affected / at risk) | 0/80 | 0/79
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Triple Therapy (MTX+SSZ+HCQ) (N=80) | TNF Inhibitor (Etanercept or Adalimumab) (N=79)
Renal Calculi (Renal and urinary disorders) | 0 (0) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myocardial Infarction (Cardiac disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Neoplasms Benign Malignant And Unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Urinary Tract Infection (Renal and urinary disorders) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-06-22): https://cdn.clinicaltrials.gov/large-docs/21/NCT02374021/Prot_000.pdf
  • Statistical Analysis Plan (2021-05-08): https://cdn.clinicaltrials.gov/large-docs/21/NCT02374021/SAP_001.pdf